CLINICAL TRIAL: NCT06228313
Title: Evaluation of Commonly Used Blood Glucose Meters in Vietnam and Effect of Hematocrit on Device's Accuracy
Brief Title: Evaluation of Commonly Used Blood Glucose Meters in Vietnam
Status: Completed | Type: Observational
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Huan Nguyen Pham, Technical supervisor, Hung Vuong Hospital
Other Study IDs: CS/HV/21/18
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy in Diabetic; Diabetes
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood sample in EDTA-NaF tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Most BGM (blood glucose monitoring) devices in Vietnam are manufactured for home use only. However, they are commonly used in healthcare facility, primarily at point of care. We want to assess the validity of these devices by using CLSI (Clinical and Laboratory Standards Institute) POCT12-A3 to assess the accuracy.

Objective: To validate the accuracy and effect of hematocrit on these devices, along with the precision profile using CLSI EP15A3

Study design: This is a cross-sectional study.

Study population: Because we need a wide range of blood glucose level. We chose pregnant women who underwent 75g glucose tolerance test.

DETAILED DESCRIPTION:
Most blood glucose monitors circulating the market are manufactured after ISO 15197:2013 standard, which is intended for self-measurement. Medical organizations need to verify blood glucose monitors if they are designed for prescription point-of-care use or validate blood glucose monitors if they are designed for over-the-counter use.

Pregnant women are selected after consent, their blood are then drawn by phlebotomist into an EDTA (ethylenediamine tetraacetic acid) with NaF (sodium flouride) blood tube. Samples are run on alinity h hematology analyzer, manufactured by Abbott, to measure hematocrit. The analyzers are verified by laboratory procedure, recommended by CLSI (Clinical and Laboratory Standards Institute) method and quality control is checked before in accordance to the laboratory procedure. After that, blood tube is mixed thoroughly before being pipetted. Each BGM device will measure blood glucose level of the pipetted whole blood. Finally, samples will be run on a cobas c 502 analyzer to measure plasma glucose level, which is a reference method for determining the accuracy of the BGM devices.

Statistical analysis: Meter performance is acceptable for use in hospitals when 95% of the individual results from the POC glucose meter system agree within 0.67 mmol/L (12 mg/dL) of the laboratory analyzer values at glucose concentrations below 5.55 mmol/L (100 mg/dL) and within 12.5% of the laboratory analyzer values at glucose concentrations at or above 5.55 mmol/L (100 mg/dL). In addition, the sum of the number of individual results with 1) errors that exceed 0.83 mmol/L (15 mg/dL) at glucose concentrations below 4.2 mmol/L (75 mg/dL) and 2) errors that exceed 20% at glucose concentrations at or above 4.2 mmol/L (75 mg/dL) should not exceed 2% of all results. An ordinary linear regression is performed to see how well the glucose level of BGM devices correlates with the reference method. Bland-Altman difference plots are used to describe the difference along with the hematocrit of each sample.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergo 75g glucose tolerance test

Exclusion Criteria:

* Usage of anticoagulant drug
* History of bleeding disorders.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women at obstetrics clinics at Hung Vuong Hospital
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Hematocrit | Each participant's blood samples are run immediately after phlebotomy
  Hematocrit in percentage, measured on hematology analyzer alinity h
Reference Glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on reference glucose analyzer cobas c 502
ACCU-CHEK Inform II glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on assessed blood glucose monitoring device ACCU-CHEK Inform II, Serial number UU14463019
ACCU-CHEK performa glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on assessed blood glucose monitoring device ACCU-CHEK performa, Serial number 68827245972
ONETOUCH VerioVue glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on assessed blood glucose monitoring device ONETOUCH VerioVue, Serial number YEPMT06H
Contour Plus glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on assessed blood glucose monitoring device Contour Plus, Serial number 6128289
EasyGlucose glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on assessed blood glucose monitoring device EasyGlucose, Serial number G16D21I0700816
VivaChek Ino glucose concentration | Each participant's blood samples are run immediately after phlebotomy
  Glucose concentration, measured on assessed blood glucose monitoring device VivaChek Ino, Serial number 311Z0021DFA

CONTACTS AND LOCATIONS:
Overall Officials: Huan N Pham, M.D., Principal Investigator — Hung Vuong Hospital
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: 3 months after publication